CLINICAL TRIAL: NCT00838188
Title: Energy Expenditure in Breast and Bottle Feeding Preterm Infants Fed Their Mother's Breast Milk
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Irit berger Dr., Tel-Aviv Sourasky Medical Center
Other Study IDs: 920060356
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Preterm Infants
Keywords: Metabolic rate; indirect calorimetry; oral feeding

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: computer-generated random numbers in sealed opaque envelopes to assign the breast/bottle sequence
  Interventions: Other: Way of Feeding - Breast feeding vs. Bottle feeding
- 2: computer-generated random numbers in sealed opaque envelopes to assign the breast/bottle sequence
  Interventions: Other: Way of Feeding - Breast feeding vs. Bottle feeding
- Breast - feeding first: computer-generated random numbers in sealed opaque envelopes to assign the breast/bottle sequence
  Interventions: Other: Way of Feeding - Breast feeding vs. Bottle feeding
- Bottle first: computer-generated random numbers in sealed opaque envelopes to assign the breast/bottle sequence
  Interventions: Other: Way of Feeding - Breast feeding vs. Bottle feeding
- Way of feeding: Each infant is evaluated twice, once after breastfeeding and once after bottle feeding of breast milk using a Premature Nipple & Ring (Ross Products Division, Columbus OH, USA). In this way, each infant serves as its own control. REE is recorded for 20 minutes after each meal
  Interventions: Other: Way of Feeding - Breast feeding vs. Bottle feeding

INTERVENTIONS:
Other: Way of Feeding - Breast feeding vs. Bottle feeding — Each infant was evaluated twice, once after breastfeeding and once after bottle feeding of breast. Computer-generated random numbers in sealed opaque envelopes to assign the breast/bottle sequence

SUMMARY:
OBJECTIVE. Neonatologists consider early feeding at the breast to be too tiring for preterm infants, although there is no evidence that this is actually the case. It is also not known whether the method of feeding affects energy expenditure. We hypothesized that resting energy expenditure (REE) would be higher after breastfeeding than after bottle feeding.

PATIENTS AND METHODS. preterm ( >32 weeks GA) stable infants who are nourished entirely by their mothers' breast milk will be studied when fed expressed breast milk either by bottle or at the breast. REE will be measured for 20 minutes after feeding. Breast milk quantity is evaluated by pre- and post feeding weighing.

DETAILED DESCRIPTION:
Most VLBW infants cannot be fed at the breast upon birth, and expressed breast milk by gastric tube is thus recommended. Sucking skills mature at around 34 weeks when nipple-feeding is introduced. In the absence of evidence-based data to decide the best timing to introduce breastfeeding, many clinicians use empiric criteria, such as the infant's weight, gestational age, and the ability of infants to bottle feed as proxies of readiness to breastfeed. Despite some evidence of physiological benefits of preterm infants feeding at the breast, many neonatologists consider direct breastfeeding to be too fatiguing for preterm infants. It is not known, however, whether preterm infants who are breastfed expend more energy than bottle-fed infants

ELIGIBILITY:
Inclusion Criteria:

* Thermally stable infants were nursed in an open and unwarmed bassinet.
* All fed solely by their mothers' breast milk equivalent to at least 150 cc/kg/day divided into eight meals and growing steadily

Exclusion Criteria:

* Infants with congenital anomalies and infants who had either more than five daily episodes of apnea of prematurity or any apnea requiring assistance or methylxanthine therapy

Ages: 34 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born after 32 weeks of gestation, when they reached the corrected gestational age of 34 weeks or more.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-11; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study was to compare resting energy expenditure (REE) in preterm infants who were fed their mothers' expressed milk by bottle and at the breast | 20 minutes after each meal

SECONDARY OUTCOMES:
Creamatocrit of the bottle at the beginning and the completion of every feeding at the breast were measured | Not relevant

CONTACTS AND LOCATIONS:
Overall Officials: Irit Berger, MD, Principal Investigator
Locations (2):
- Israel (2):
  - Department of Neonatology, Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Berger I, Weintraub V, Dollberg S, Kopolovitz R, Mandel D. Energy expenditure for breastfeeding and bottle-feeding preterm infants. Pediatrics. 2009 Dec;124(6):e1149-52. doi: 10.1542/peds.2009-0165. Epub 2009 Nov 23. PMID 19933725